CLINICAL TRIAL: NCT00512304
Title: Feasibility Study of 2 Parallel Phases II Pre or Postgastrectomy in Patients With Gastric Cancer (FOLFIRI-radiotherapy Plus 5 Fluorouracil-surgery or Surgery-FOLFIRI-radiotherapy Plus 5 Fluorouracil)
Brief Title: Adjuvant Treatment of Gastric Cancer With Chemotherapy and Chemoradiotherapy (TRACE)
Acronym: TRACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/097/HP
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preoperative chemoradiotherapy (Experimental)
  Interventions: Procedure: association chemotherapy and radiochemotherapy
- Postoperative chemoradiotherapy (Experimental)
  Interventions: Procedure: association chemotherapy and radiochemotherapy

INTERVENTIONS:
Procedure: association chemotherapy and radiochemotherapy

SUMMARY:
Post-operative radio-chemotherapy decrease the recurrence risk of gastric cancer(N Engl J Med 2001). However the chemotherapy regimen (5 fluorouracil IV bolus) used was toxic and suboptimal. We propose to evaluate in adjuvant situation an active and well tolerate chemotherapy regimen (FOLFIRI)in patients with metastatic gastric cancer. During the radiotherapy we will use 5 FU continue infusion as previously reported. The global design of adjuvant treatment will be four FOLFIRI courses, radiotherapy (45 Gy)with 5FU IV continue then four FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma histologically confirmed
* tumor T3 or N+ at the pretherapeutic staging (Scanner and endoscopic ultrasound)
* performance status WHO<2
* serum albumin >30 gr/l
* weight loss < 10% in the next 6 months
* signed informed consent form

Exclusion Criteria:

* metastatic disease
* prior abdominal radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
feasibility of treatment | at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL Pierre, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University hospital, Rouen, France